CLINICAL TRIAL: NCT02833545
Title: Safety and Efficacy of Intra-articular Ozone Injections for Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, DROR ROBINSON, Head Orthopedic Research Unit, Rabin Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 751-15-RMC
Record Dates: First submitted 2016-06-19; First posted 2016-07-14 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Osteoarthritis Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Steroids

STUDY DESIGN:
Intervention Model Description: A sequential series of patients receiving steroid injections was compared to a sequential series of patients receiving ozone injections
Who Masked: Investigator, Outcomes Assessor
Masking Description: the outcome assessor was not aware of the therapy administered
Oversight: Data Monitoring Committee: No

ARMS (2):
- OZONE (Experimental): injection of ozone gas
  Interventions: Device: Ozone gas
- control (Active Comparator): injeciton of steroids intra articularly
  Interventions: Drug: Steroid injection

INTERVENTIONS:
Device: Ozone gas — Injection of ozone gas intra articularly
  Arms: OZONE
Drug: Steroid injection — Injection of steroids (diprospan) intra articularly
  Arms: control

SUMMARY:
Prospective, Interventional, Non-Randomized, Open Label, Single Group Assignment, Single Center.

ELIGIBILITY:
Inclusion Criteria:

* 55 to 79 years of age
* Symptomatic Knee osteoarthritis
* VAS pain intensity is at least 40 mm on a 100 mm scale
* Must be physically and mentally willing and able to comply with post-operative rehabilitation and routinely schedule clinical and radiographic visits.

Exclusion Criteria:

* Any known tumor of the ipsilateral knee.
* Any known infection of the treated knee.
* Osteoarthritis of the operated knee Kelgren Lawrence < grade 2.
* Chemotherapy treatment in the past 12 months.
* Patients who are sensitive to ozone.
* Pregnant women, or breastfeeding women.
* Evidence of any significant systemic disease (such as but not limited to HIV infection, hepatitis infection or HTLV infection), known coagulopathies, that might compromise the Subject's welfare.
* Substance abuse or alcohol abuse.
* Participation in other clinical trials in parallel to this study.

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Improvement in VAS Pain intensity | 6 months
  The outcome measure will be measured according to patient response to the question: during the last week what was your average pain intensity. The response will be measured in millimeters as marked on a 10 cm long line. No pain equals 0 mm and maximal possible pain equals 100mm